CLINICAL TRIAL: NCT06330415
Title: Web-based Intervention Supporting Employers of Small and Medium-sized Enterprises During the Return to Work of Employees on Long-term Sick-leave: Design of a Randomised Controlled Trial
Brief Title: Effect and Process Evaluation of the SME Tool
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Frederieke Schaafsma, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25603
Record Dates: First submitted 2024-02-14; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Sick-listed Employees

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Unlimited access to the SME tool.
  Interventions: Other: The SME tool
- Control group (No Intervention): Care as usual by the occupational health service.

INTERVENTIONS:
Other: The SME tool — The intervention comprises of an open-access website targeting the employer of the sick-listed employee. The website provides practical resources, including templates, communication videos and information on legislation, workplace accommodations and most common reasons of sickness absence.
  Arms: Intervention group

SUMMARY:
A web-based tool has been developed to help small and medium-sized businesses support employees returning to work after sick-leave. A six-month trial is conducted, randomly assigning employer-employee dyads to either use the tool or receive standard care. The primary aim is to evaluate its impact on employee satisfaction with return-to-work support.

ELIGIBILITY:
Inclusion Criteria:

Employees at study enrolment should:

* be of working age (18-65 years);
* have a fixed or temporary employment contract at a SME (≤ 250 employees), with a minimum of 6 months remaining in their contract;
* be currently sick-listed or partially sick-listed (≤8 weeks), with a risk of long-term absenteeism, based on the likelihood of the duration of sickness absence exceeding two months as assessed by their occupational physician;
* be able to understand and read Dutch sufficiently, in order to complete the questionnaires.

The employer of the participating employee will be included. At time of study entry, the employer should be:

* an employer, supervisor, (case)manager or HR manager of a SME (≤ 250 employees). In this study, the employer is appointed by the employee and refers to the person who is the direct supervisor, in direct contact with the employee, and thus the person who offers the RTW support to the employee;
* able to understand and read Dutch sufficiently, in order to use the intervention and complete the questionnaires.

Exclusion Criteria:

• Not have a colleague who is already participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with the RTW support of employer assessed by the employee | Baseline (T0), 1 month (T1), 3 month (T2) and 6 month (T3) follow-up
  The primary outcome is the employee satisfaction regarding the return-to-work support provided by the employer. This is measured using a single-item rating in a questionnaire: 'How satisfied are you with the sick-leave and return to work guidance you have received from your employer since the sick-leave/over the past month/3 months?', graded on a 5-point Likert scale ranging from very dissatisfied to very satisfied. The numerical scores assigned reflect the level of satisfaction, with higher scores indicative of higher satisfaction.

SECONDARY OUTCOMES:
Social support | Baseline (T0), 1 month (T1), 3 month (T2) and 6 month (T3) follow-up
  Social support is assessed through the four aspects of support, i.e.: 1) emotional support, 2) practical support, 3) informational support, and 4) appreciative support. The assessment entails eight questions in a questionnaire that inquire the importance and amount of support received, for example: 'How important is it that your employer provides emotional support during sick-leave and RTW? Explanation: Emotional support refers to the degree, we to which the employer shows understanding and listens to your concerns.' Response categories are: 1) very unimportant, 2) unimportant, 3) neutral, 4) important, and 5) very important. The mean score of the total sum is calculated, with higher scores indicating higher social support from the employer, collectively evaluating the overall level of social support provided by the employer.
Total number of sick-leave days | Baseline (T0), 1 month (T1), 3 month (T2) and 6 month (T3) follow-up
  The total number of sick-leave days involves the assessment of the average number of working hours per week over the preceding four weeks and the total number of (partial) sick days, measured in a questionnaire. Answer categories include yes or no options and open-ended responses to express current employment status, for example date input (e.g., return to work since: ../../….).
Work performance | Baseline (T0), 1 month (T1), 3 month (T2) and 6 month (T3) follow-up
  Work performance is evaluated using scale 2A from the Maastricht Instrument for Sustainable Employability (MAISE), reflecting the long-term capacity of employees to actively engage in and contribute to the workforce. The scale consists of six statements in a questionnaire, to be completed only if work tasks have been done in the past four weeks. For example: 'I have the knowledge to perform my job well.', are measured on a 5-point Likert scale. Response categories are: 1) completely disagree, 2) disagree, 3) neutral, 4) agree, and 5) completely agree. The mean score is calculated, with higher scores indicating higher work performance.
Quality of working Life | Baseline (T0), 1 month (T1), 3 month (T2) and 6 month (T3) follow-up
  Quality of Working Life is measured using the Quality of Working Life Questionnaire for cancer survivors (QWLQ-CS). Subscale 2 about understanding and recognition in the organization, consisting of 5 items, is included in the questionnaire. For example: 'My supervisor understands my health situation and possible complaints.', measured on a 6-point Likert scale. Response categories comprise: 1) completely disagree, 2) disagree, 3) somewhat disagree, 4) somewhat agree, 5) agree, and 6) completely agree. The sum represents the overall score, with a higher score corresponding to a higher quality of working life.
Self-efficacy | Baseline (T0), 1 month (T1), 3 month (T2) and 6 month (T3) follow-up
  Self-efficacy pertains to the perceived capability of the employer to effectively support employees during sickness absence. This evaluation is conducted with three items concerning meaningfulness, impact and skills, of the competence scale of the Empowerment Questionnaire. For example, statements such as: 'Supporting an employee who has reported sick is a significant responsibility for me.', are measured in a questionnaire on a 6-point Likert scale. Response categories are: 1) completely disagree, 2) disagree, 3) somewhat disagree, 4) somewhat agree, 5) agree, and 6) completely agree. The mean score of the sum is calculated, with higher scores reflect higher self-efficacy.
Satisfaction with the resumption of work of the respective employee | Baseline (T0), 1 month (T1), 3 month (T2) and 6 month (T3) follow-up
  Satisfaction with the resumption of work of the respective employee: This is measured with one self-developed question in a questionnaire: 'How satisfied are you with the work resumption process of your employee in the past month/3 months?', on a 5-point Likert scale. Response categories are: 1) very dissatisfied, 2) dissatisfied, 3) neutral, 4) satisfied, and 5) very satisfied. The category represents the overall score, with a higher score reflecting higher satisfaction.

OTHER OUTCOMES:
Recruitment | 1 month (T1), 3 month (T2) and 6 month (T3) follow-up
  For the process evaluation, recruitment is measured through reasons for non-participation and the usefulness of recruitment strategies. This is measured in CASTOR with an open ended question, filled in by recruited employees who wish to not participate prior to the trial. Also a logbook related to recruitment strategies is maintained by the researchers, containing details about what recruitment strategy is used during the trial and the corresponding outcome.
Use of the SME tool | 3 month (T2) and 6 month (T3) follow-up
  For the process evaluation, the use of the SME tool is measured with questions regarding number of visits, duration of visits, tool availability and web analytics. For example with the question: 'How often have you visited the SME tool in the past three months?'. Response categories comprise multiple choice and open ended options.
Perceived usefulness of the SME tool | 3 month (T2) and 6 month (T3) follow-up
  For the process evaluation, the perceived usefulness of the SME tool is measured with self-developed questions regarding the usefulness of the tool, enhancement of knowledge and skills, and likelihood of recommending the tool to colleagues. For example through the question: 'Would you recommend the tool to other employers when guiding an employee who has reported ill?'. Response categories are multiple choice and open ended options.
Components of the logic model of change | 1 month (T1), 3 month (T2) and 6 month (T3) follow-up
  For the process evaluation, the logic model of change components consists of the constructs: autonomy, competence, relatedness and ability. These are measured in self-developed questions such as: 'I have the skills to support an employee on sick leave.', measured on a 6-point Likert scale. Response categories comprise: 1) completely disagree, 2) disagree, 3) somewhat disagree, 4) somewhat agree, 5) agree, and 6) completely agree. Individual scores represent the overall score of individual component, with higher score reflecting higher autonomy, competence, relatedness and ability.
Experiences | Cross-sectional after 6 months follow-up
  For the process evaluation, the interpretation of the results from the RCT and potential implementation strategies for the national implementation of the tool will be explored via one-time interviews with 5-10 employees, 5-10 employers, and 5-10 OPs, out of a purposive sample of RCT participants.

CONTACTS AND LOCATIONS:
Overall Officials: Frederieke Schaafsma, Prof. dr., Principal Investigator — Amsterdam UMC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beerda DCE, Greidanus MA, de Rijk AE, de Wind A, Tamminga SJ, Schaafsma FG. The SME tool supporting employers of small- and medium-sized enterprises during the return to work of employees on long-term sick leave: study protocol for a randomized controlled trial and for a process evaluation. Trials. 2024 Aug 16;25(1):541. doi: 10.1186/s13063-024-08383-4. PMID 39152487